CLINICAL TRIAL: NCT00912249
Title: The Clinical Application of Horticulture Therapy in Psychiatric Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 098019-3
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-04

CONDITIONS: Horticulture Therapy in Psychiatric Rehabilitation
Keywords: Horticulture Therapy; Psychiatric Rehabilitation; Nature-assisted psychotherapy; Day Care
MeSH Terms: interventions — Horticultural Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Horticultural Therapy (Experimental)
  Interventions: Behavioral: Horticulture Therapy

INTERVENTIONS:
Behavioral: Horticulture Therapy — We will design courses of Horticultural therapy to provide to the Patients in Day Care Unit

SUMMARY:
Horticultural Therapy (HT) uses plants, gardening, and the close relationship between well-beings and plants. It integrates effort, hope, expectation, harvest and the enjoyment of whole process to help people with disabilities. During the process, patient can learn more about themselves and experience the nature.

It can be traced to 1798, Dr. B. Rush found farm work helped people with mental illness. Today, horticulture therapy is well applied in disabilities, elderly and children. It needs detailed evaluation for the condition of illness to achieve optimal efficacy. It contains two parts- to sense and to operate! Patients can relax themselves and learn to work with others, realize the responsibility of caring another life, understand their relationship with environment. Patient can tolerate frustration better via acceptance the withered plants. In cultivation, it trains patient the occupational technique ( to operate instrument), communication, social skill, independence, stable mood.

Based on studies, 0ne third patients with mental illness stabilized after treatment. However, aggressive rehabilitation is necessary to maintain their function. In our study, it plans to incorporate horticulture therapy into psychiatric clinical practice in our hospital. We plan to recruit horticulture therapist, visiting staffs, residents, occupational therapists and nurses to participate the design and operation in class.

This program will recruit patients with schizophrenia, bipolar disorder, organic brain syndrome and other mental illness in our daycare. We will help patients with personal treatment record. We will use case study to report some typical cases. All the cases will be investigated qualitatively with intensive interview to explore the subjective experience on this therapy. We will also use simple questionnaire to found quantitative study in the further.

To sum up, this program helps the connection for horticulture therapy and psychiatric rehabilitation. It promotes " patient-centered" support and offers physical, mental , social, spiritual services. It not only produces academic performance but fulfills the ideal of holistic health care!

ELIGIBILITY:
Inclusion Criteria:

* 18~65 both sexes
* Adequate daily function for horticultural activities
* Day care patients or referred from OPD
* Willing to accept and cooperate with H/T

Exclusion Criteria:

* Substance abuser or PD
* Severe suicide or harmful behaviors
* Severe physical problem impeding horticultural activities
* Lack of motivation for H/T

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview and Questionnaire for satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chun-lin Chen, MD, MA, Study Director — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taiwan